CLINICAL TRIAL: NCT07299162
Title: The Effect of Virtual Reality Therapy on Upper Extremity Functions in Subacute Stroke Patients Receiving Conventional Rehabilitation and Action Observation Therapy: A Randomized Controlled Single-Blind Study
Brief Title: The Effect of Virtual Reality Therapy on Upper Extremity Functions in Subacute Stroke Patients Receiving Rehabilitation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Physical Medicine Rehabilitation Training and Research Hospital (Other Government)
Collaborators: Inosens information technologies limited company (Unknown)
Responsible Party: Principal Investigator, Seda Akbayrak, Resident Doctor, Istanbul Physical Medicine Rehabilitation Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2025-32
Record Dates: First submitted 2025-11-25; First posted 2025-12-23 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2025-11

CONDITIONS: Stroke; Hemiplegia and/or Hemiparesis Following Stroke
Keywords: Virtual reality; action observation therapy; hemiplegia; hemiparesis; stroke; upper extremity
MeSH Terms: conditions — Stroke; Hemiplegia; Paresis | interventions — Exergaming; Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual Reality (Active Comparator): Patients in this group will receive virtual reality rehabilitation for 5 weeks, 3 times a week for a total of 15 sessions. Additionally they will receive conventional rehabilitation six days a week for 5 weeks and action observation therapy for 3 times a week for 5 weeks. For action observation therapy 1 session each week will be done under supervision of principal investigator and 2 sessions will performed independently by the patient
  Interventions: Other: Virtual Reality; Other: Conventional rehabilitation; Other: Action observation therapy
- Control (Other): Patients in this group will receive conventional rehabilitation six days a week for 5 weeks and action observation therapy for 3 times a week for 5 weeks. For action observation therapy 1 session each week will be done under supervision of principal investigator and 2 sessions will performed independently by the patient
  Interventions: Other: Conventional rehabilitation; Other: Action observation therapy

INTERVENTIONS:
Other: Virtual Reality — Camera controlled virtual reality games for upper extremity
  Other Names: exergame
  Arms: Virtual Reality
Other: Conventional rehabilitation — Personalized conventional exercises for hemiparesis after stroke
  Other Names: exercise
Other: Action observation therapy — Rehabilitation method that involves patients watching video recordings of purposeful upper extremity movements designed for daily life activities followed by physically attempting the same movements.

SUMMARY:
Stroke ranks second among the leading causes of death worldwide and third among the causes of disability. In stroke patients, motor impairment typically affects facial movements and the upper and lower extremities unilaterally. Upper extremity involvement, in particular, negatively impacts patients' activities of daily living, such as eating and dressing. Various rehabilitation methods are used to improve the function of the paretic upper extremity in stroke patients. Action Observation Therapy and Virtual Reality are among the rehabilitation approaches currently used to support upper extremity rehabilitation.

In our study, patients will be randomly divided into two groups: one group will receive conventional rehabilitation and Action Observation Therapy, while the other group will additionally receive Virtual Reality therapy. This study aims to investigate the contribution of Virtual Reality therapy, when added to conventional rehabilitation and Action Observation Therapy, to the recovery of the paretic upper extremity in patients with subacute stroke.

DETAILED DESCRIPTION:
Methodology

All volunteer patients will be evaluated at the beginning of the treatment using the following assessment tools: Fugl-Meyer Assessment-Upper Extremity, Brunnstrom Stages-Upper Extremity/Hand, Wolf Motor Function Test, Motricity Index-Arm, Stroke Impact Scale 3.0, and Task-Based Exercises (number of times the patient can bring their hand to the mouth, behind the head, and to the sacrum in one minute).

Patients will be randomly assigned to two groups using computerized randomization.

One group will receive conventional therapy 5 days per week plus Action Observation Therapy (AOT) 3 times per week for 30 minutes.

Each AOT session will consist of videos featuring goal-oriented tasks prepared according to the individual needs of the patient. The videos will change weekly. The first session each week will be supervised by the physician, while the other two sessions will be performed independently by the patient.

In AOT, each task is broken down into subcomponents. Each sub-task will be observed for 3 minutes, followed by a 2-minute practice period. For example, the task of drinking water from a glass will be divided into three sub-actions: (1) fill the glass, (2) hold the glass, and (3) bring the glass to the mouth. Each sub-action will be presented as a video for 3 minutes, followed by 2 minutes of attempted execution by the patient.

The second group will receive conventional therapy 5 days per week, plus Action Observation Therapy (as described above) and Virtual Reality therapy (exergaming) using Becure SmartPose games, 3 times per week for 30 minutes.

After completing the 5-week treatment program, a follow-up assessment will be performed at the end of treatment and one month after treatment completion.

Sample Size Calculation

The primary outcome measure is the Fugl-Meyer Assessment-Upper Extremity. Measurements will be taken at baseline, post-treatment, and one month after treatment for both the virtual reality group and the control group.

Using a medium effect size (partial eta-squared = 0.06) for repeated measures mixed model ANOVA, with α = 0.05 and power = 0.85, the minimum required sample size was calculated as 16 participants per group, 32 in total. Considering an estimated 15% dropout rate, the final sample size was adjusted to 38 participants. The calculation was performed using G*Power version 3.1.9.4 (Franz Faul, Universität Kiel, Germany).

Statistical Analysis

The normality of the data distribution will be tested using the Shapiro-Wilk test.

If data are normally distributed, repeated measures ANOVA will be used to compare all variables (Fugl-Meyer Upper Extremity, Brunnstrom Upper Extremity/Hand, Wolf Motor Function Test, Motricity Index-Arm, Stroke Impact Scale 3.0, and Task-Based Exercises).

If the overall ANOVA reveals significance (p < 0.05), Post Hoc pairwise comparisons will be conducted to determine which time points differ.

If data are not normally distributed, within-group comparisons will be conducted using the Friedman test and Wilcoxon signed-rank test, while between-group comparisons will be performed using the Mann-Whitney U test.

Bonferroni-corrected p-values < 0.05 will be considered statistically significant in post hoc comparisons.

All analyses will be conducted using SPSS version 18.0.

ELIGIBILITY:
Inclusion Criteria:

* Patients over the age of 18
* Patients in the subacute phase of stroke (between 6 weeks and 6 months post-stroke)
* Patients with a first-ever stroke
* Brunnstrom stage 3 or above for both upper extremity and hand
* Mini-Mental State Examination (MMSE) score >=20

No major medical condition that would prevent participation in the treatment

Exclusion Criteria:

* Presence of pain in the paretic shoulder severe enough to prevent exercise
* History of bilateral stroke
* Patients with global aphasia and/or cognitive impairment that significantly affects treatment compliance
* Patients with severe visual impairment
* Presence of unilateral spatial neglect
* Inability to maintain sitting balance
* Modified Ashworth Scale > 4 in the hemiplegic arm

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Estimated)
Dates: Start 2025-08-15 (Actual); Primary Completion 2026-03-25 (Estimated); Study Completion 2026-04-20 (Estimated)

PRIMARY OUTCOMES:
Fugl-Meyer Upper Extremity | From enrollment to the 1 months after treatment
  The Fugl-Meyer Assessment for Upper Extremity (FMA-UE) is a standardized scale used to assess motor recovery of the upper limb in post-stroke patients. It evaluates voluntary movement, reflex activity, coordination, and speed. The scale consists of 33 items, and the total score ranges from 0 to 66, with 0 indicating no motor function and 66 representing normal motor function. A Turkish validity and reliability study has also been conducted for this scale.

SECONDARY OUTCOMES:
WOLF motor function test - Functional Ability Scale | From enrollment to the 1 month after treatment
  The Wolf Motor Function Test (WMFT) is an assessment tool developed to evaluate motor skills in patients with upper extremity motor deficits. The test consists of 17 items. For 15 items, data is collected on functional ability and performance time, while 2 items assess muscle strength. 2 tests for muscle strength were not used.Each activity is scored on a Functional Ability Scale ranging from 0 to 5, where 0 indicates no use of the affected limb during the activity, and 5 represents normal movement. An average score is calculated for the Functional Ability Scale, with higher scores indicating better motor function.
  A Turkish version of the WMFT has also been validated and found reliable for use in stroke patients.
Motricity Index - Upper Extremity | From enrollment to the 1 month after treatment
  The Motricity Index is a scale used to determine patients' motor function levels. In our study, the Motricity Index - Upper Extremity score will be calculated to evaluate upper limb function following stroke. The minimum score is 0 and the maximum score is 99. A Turkish version of the motricity index has been validated and found reliable for use.
Stroke Impact Scale 3.0: | From enrollment to the 1 month after treatment
  The Stroke Impact Scale is a stroke-specific health status measure designed to assess the quality of life and functional independence of patients after stroke. It allows both patients and their caregivers to evaluate the patient's overall condition. The assessment uses a 5-point Likert scale for scoring. Scores for each domain range from 0 to 100. In addition to questions across 8 subdomains, SIS 3.0 includes a visual analog scale to measure perceived recovery after stroke, scored from 0 to 100 (0 = no recovery, 100 = full recovery).
Brunnstrom Upper Extremity and Hand | From enrollment to the 1 month after treatment
  The Brunnstrom method evaluates motor recovery in stroke patients through six sequential stages. Stage 1 represents the worst condition, characterized by flaccidity and no voluntary movement in the upper extremity. Stage 6 indicates the best outcome, where coordinated, voluntary, and normal movement patterns are fully restored. This scale helps clinicians determine the patient's current recovery stage and plan appropriate rehabilitation strategies.
Task Specific Exercises | From enrollment to the 1 month after treatment
  Task-specific exercises include counting how many times the patient can bring their hand to their mouth, behind their head, and to their sacrum within one minute. A higher number of repetitions within the one-minute interval indicates better upper extremity motor function.
The Wolf Motor Function Test (WMFT)- Performance Time | From enrollment to the 1 month after treatment
  The Wolf Motor Function Test (WMFT) is an assessment tool developed to evaluate motor skills in patients with upper extremity motor deficits. The test consists of 17 items. For 15 items, data is collected on functional ability and performance time, while 2 items assess muscle strength. 2 tests for muscle strength were not used. Performance Time is recorded in seconds. The maximum allowed time to complete an activity is 120 seconds. If the patient is unable to complete the activity within this time, a score of 120 seconds is assigned. Therefore, the median score is calculated for Performance Time.
  A Turkish version of the WMFT has also been validated and found reliable for use in stroke patients.

CONTACTS AND LOCATIONS:
Overall Officials: Seda Akbayrak, MD, Principal Investigator — Istanbul Physical Therapy and Rehabilitation Training and Research Hospital
Locations (1):
- Istanbul Physical Therapy and Rehabilitation Training and Research Hospital, Istanbul, Bahçelievler, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Ikbali Afsar S, Mirzayev I, Umit Yemisci O, Cosar Saracgil SN. Virtual Reality in Upper Extremity Rehabilitation of Stroke Patients: A Randomized Controlled Trial. J Stroke Cerebrovasc Dis. 2018 Dec;27(12):3473-3478. doi: 10.1016/j.jstrokecerebrovasdis.2018.08.007. Epub 2018 Sep 5. PMID 30193810
- [Result] Chen J, Or CK, Chen T. Effectiveness of Using Virtual Reality-Supported Exercise Therapy for Upper Extremity Motor Rehabilitation in Patients With Stroke: Systematic Review and Meta-analysis of Randomized Controlled Trials. J Med Internet Res. 2022 Jun 20;24(6):e24111. doi: 10.2196/24111. PMID 35723907
- [Result] Yu JA, Park J. The effect of first-person perspective action observation training on upper extremity function and activity of daily living of chronic stroke patients. Brain Behav. 2022 May;12(5):e2565. doi: 10.1002/brb3.2565. Epub 2022 Apr 10. PMID 35398981
- [Result] Pollock A, Farmer SE, Brady MC, Langhorne P, Mead GE, Mehrholz J, van Wijck F. Interventions for improving upper limb function after stroke. Cochrane Database Syst Rev. 2014 Nov 12;2014(11):CD010820. doi: 10.1002/14651858.CD010820.pub2. PMID 25387001